CLINICAL TRIAL: NCT02294279
Title: The Evaluation of FeNO for Predicting Response to an Inhaled Corticosteroid in Subjects With Non-specific Respiratory Symptoms
Brief Title: The Evaluation of FeNO for Predicting Response to ICS in Subjects With Non-specific Respiratory Symptoms
Acronym: NSRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OR01013
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: cough, wheeze, dyspnoea
MeSH Terms: conditions — Asthma; Cough; Respiratory Sounds; Dyspnea | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): 4 weeks of corticosteroid treatment with QVAR (100mcg), 400 mcg daily; two puffs twice daily
  Interventions: Drug: Qvar (100 mcg)
- Placebo (No Intervention): Blinded placebo inhaler

INTERVENTIONS:
Drug: Qvar (100 mcg) — 2 puffs twice daily; 400 mcg daily over 4 weeks treatment period
  Other Names: Beclomethasone diproprionate
  Arms: Active

SUMMARY:
Nitric Oxide is recognized as a biological marker for many chronic airway diseases. It has been standardised for clinical use indicating airway inflammation.

In clinical practice, FeNO can aid confirmation of an asthma diagnosis and can indicate the degree of steroid-responsiveness. This can help guide physician decisions on the initiation of inhaled corticosteroid (ICS) therapy, or adjustment of ICS therapy.

Therefore, FeNO measurement could be particularly useful to confirm an asthma diagnosis in patients with non-specific respiratory symptoms (≥ 6 weeks of cough and/or wheezing and/or chronic dyspnoea) and to assess how likely they are to benefit from corticosteroid treatment.

This study will assess the suitability of FeNO to predict ICS responsiveness in patients with non-specific respiratory symptoms.

Additionally, we would like to determine the suitability of FeNO as a diagnostic tool for asthma in comparison to conventional predictors, e.g. spirometry.

DETAILED DESCRIPTION:
Randomised, double-blind, placebo-controlled trial with planned enrolment of 264 patients from the UK and Singapore. Eligible patients are 18-80 years old with ≥6 weeks' duration of non-specific respiratory symptoms defined as cough and/or wheeze and/or dyspnoea. Patients with FEV1 <90% predicted at visit 1 must show reversibility of <20% at visit 1 or within the prior year. Key exclusion criteria are prior diagnosis of asthma; evidence of concomitant chronic respiratory disease, respiratory tract infection; or known significant risk factor for cough or wheeze.

Baseline assessments will include spirometry (FEV1, forced vital capacity) and FeNO measurement. Patients will be provided with a peak flow meter for twice daily measurement throughout the study. At 2 weeks, a clinical assessment and spirometry will be performed to confirm eligibility, and patients will complete four validated questionnaires to assess quality of life, asthma control, and asthma symptoms, including a visual analog scale for bother from asthma symptoms. Eligible patients will then be stratified by baseline FeNO level (normal ≤25, intermediate >25 to ≤50, or high >50 ppb); each group will be randomised to receive beclometasone 400 mcg daily or placebo for 6 weeks. An optional blood sample will be collected from consenting patients to assess blood eosinophils.

At visit 3, final assessments will include spirometry, FeNO measurement, and all questionnaires. Interaction analysis will be used to determine whether a differential effect exists in response to ICS between FeNO groups.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained before conducting any study-related procedures
* The patient is a man or woman aged 18 to 80 years as of the screening visit
* The patient is experiencing non-specific respiratory symptoms defined as follows: Cough and/or wheeze and/or chronic dyspnoea for ≥ 6 weeks prior to visit 1
* Patients displaying an FEV1< 90% predicted at visit 1, will also need to show a reversibility to a short-acting beta-agonist of < 20% at visit 1 or within the previous year
* Women of childbearing potential (post-menarche or less than 2 years post-menopausal or not surgically sterile) must be willing to commit to using a medically accepted method of contraception for the duration of the study. Accepted methods of contraception include: intrauterine devices (IUD), systemic contraception e.g. steroidal contraceptives (oral, implanted transdermal or injected), barrier methods with spermicide, and partner vasectomy

Exclusion Criteria:

* The patient has ever been diagnosed with asthma as evidenced by the UK quality outcome framework approved Read code as well as a reversibility of ≥ 20% predicted
* The patient has received oral, inhaled or systemic corticosteroids, a leukotriene modifier or long-acting-beta-agonist within four weeks prior to visit 1. All therapy and treatment other than those outlined are permitted during the study
* The patient has a significant chronic respiratory disorder other than asthma, e.g. COPD (fixed obstruction, post-bronchodilator) cystic fibrosis, severe and untreated bronchiectasis or interstitial lung disease
* The patient has a significant medical condition that would make it unlikely for the patient to complete the study
* The patient has a known significant risk factor for cough or wheeze, including but not limited to: taking an ACE inhibitor, severe untreated rhinitis, or significant gastroesophageal reflux disease
* The patient is asymptomatic (ACQ < 1) after the initial 2-week assessment
* The patient has had a respiratory tract infection as judged clinically, within four weeks prior to visit 1, or displays an acute respiratory tract infection at the time of the study
* The patient is a pregnant woman or intends to get pregnant (Any woman becoming pregnant during the study will be withdrawn from the study)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | Baseline and 4 weeks
  The Asthma control questionnaire (ACQ) is a seven question (i.e. the top scoring 5 symptoms, daily rescue bronchodilator use and FEV1% pred.), validated tool for assessing asthma control. Patients are asked to recall how their asthma has been during the last 7 days and to evaluate their asthma against 5 symptom questions and a rescue bronchodilator use question on a 6-point scale (0 = no impairment, 6 = maximum impairment). In addition, the research nurse will grade the FEV1 % predicted on a 6 point scale (0 to 6). The questions are equally weighted and ACQ7 score is the mean of the 7 questions, generating a value between 0 (totally controlled) and 6 (severely uncontrolled).

SECONDARY OUTCOMES:
EuroQol 5 dimension questionnaire | Baseline and 4 weeks
  The EQ-5D-3L questionnaire is a validated instrument that derives a person's health profile. The EQ-5D-3L consists of two parts. The first one is the EQ descriptive system which comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The respondent is asked to indicate their health state by ticking the most appropriate statement (no problems to extreme problems). The second part is the EQ visual analog scale (EQ VAS). It records the respondent's self-rated health on a 20 cm vertical,visual analogue scale with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Visual Analogue Scale test (VAS) and cough Visual analogue scale test | Baseline and 4 weeks
  Patients rate their symptom/cough severity by placing a mark on a line to indicate symptom severity.
Spirometry (PEF, FEV1, FVC, FEV1/FVC) | 3 days
  Spirometry will be conducted to obtain an objective measure of the patient's lung function
Eosinophil analysis | 1 day
  A blood test will be taken from consenting patients to assess the eosinophil level as marker for inflammation.
Peak expiratory flow (PEF diary) | From visit 1 till 6 weeks follow-up (2 recordings per day over 6 weeks)
  Peak expiratory flow will be measured using a portable peak flow meter.
Global Evaluation of Treatment Effectiveness Scale (GETE) | 1 day
  Clinical judgment on whether the treatment was successful on a 5-point scale

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof, Study Director — Research in Real Life
Locations (1):
- Research in Real Life Ltd, Oakington, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Principal investigator has not made a decision regarding a plan to share data at this point in time.

REFERENCES:
- [Derived] Price DB, Buhl R, Chan A, Freeman D, Gardener E, Godley C, Gruffydd-Jones K, McGarvey L, Ohta K, Ryan D, Syk J, Tan NC, Tan T, Thomas M, Yang S, Konduru PR, Ngantcha M, d'Alcontres MS, Lapperre TS. Fractional exhaled nitric oxide as a predictor of response to inhaled corticosteroids in patients with non-specific respiratory symptoms and insignificant bronchodilator reversibility: a randomised controlled trial. Lancet Respir Med. 2018 Jan;6(1):29-39. doi: 10.1016/S2213-2600(17)30424-1. Epub 2017 Nov 3. PMID 29108938